CLINICAL TRIAL: NCT05162937
Title: A Randomized, Double-blind, Placebo-controlled Clinical Trial to Evaluate the Preliminary Efficacy, Safety, Pharmacokinetics and Immunogenicity Characteristics of GR1501 Injection by in Patients With Active Axial Spondyloarthritis
Brief Title: to Evaluate the Preliminary Efficacy and Safety of GR1501 Injection in Patients With Active Axial Spondyloarthritis
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Genrix (Shanghai) Biopharmaceutical Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: GR1501-002
Record Dates: First submitted 2021-09-17; First posted 2021-12-20 (Actual); Last update posted 2023-04-05 (Actual); Status verified 2023-04

CONDITIONS: Axial Spondyloarthritis
Keywords: IL-17A; Axial Spondyloarthritis
MeSH Terms: conditions — Axial Spondyloarthritis

STUDY DESIGN:
Intervention Model Description: A total of 160 patients were enrolled in the planned trial, and after passing the screening period of 2 weeks, they were randomly assigned to the 100mg group, 200mg group, 300mg group or placebo group according to 1:1:1:1. After the completion of the 16-week administration period, the follow-up period (~24 weeks) was initiated.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Double blind
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Treatment group 1 (Experimental): Drug：GR1501 100mg
  Interventions: Biological: IL-17A antibody
- Treatment group 2 (Experimental): Drug：GR1501 200mg
  Interventions: Biological: IL-17A antibody
- Treatment group 3 (Experimental): Drug：GR1501 300mg
  Interventions: Biological: IL-17A antibody
- Treatment group 4 (Placebo Comparator): Drug：placebo
  Interventions: Biological: IL-17A antibody

INTERVENTIONS:
Biological: IL-17A antibody — Recombinant fully human IgG4 anti-IL-17A monoclonal antibody drug

SUMMARY:
Dosage: 100mg or 200mg or 300mg Administration frequency: Q2W administration in the first 4 weeks (W0, W2, W4), and subsequent Q4W administration (W8, W12) Administration: subcutaneous injection Specifications: 100mg/ 1mL/bottle or placebo 0mg/1ml/ bottle

DETAILED DESCRIPTION:
This is a randomized, double-blind, placebo-controlled phase II clinical trial evaluating the preliminary efficacy, safety, pharmacokinetic, and immunogenicity of GR1501 injection (IL-17A antiboby) at different doses and dosing frequency in patients with active axial spinal arthritis.

A total of 160 patients were enrolled in the planned trial, and after passing the screening period of 2 weeks, they were randomly assigned to the 100mg group, 200mg group, 300mg group or placebo group according to 1:1:1:1.After the completion of the 16-week administration period, the follow-up period (~24 weeks) was initiated.

ELIGIBILITY:
Inclusion Criteria:

1. According with the diagnosis of axial spondyloarthritis (axSpA) by the Assessment of Spondyloarthritis International Society (ASAS);,
2. During the screening period, the Bath Ankylosing Spondylitis Disease Activity Index (BASDAI) ≥ 4 points and the Spinal Pain (BASDAI Article 2) NRS score ≥ 4 points;

Exclusion Criteria:

1. Previous or current Crohn's disease;
2. Suffering from ulcerative enteritis and requiring immunosuppressive therapy at present;

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 160 (Actual)
Dates: Start 2020-09-07 (Actual); Primary Completion 2021-07-30 (Actual); Study Completion 2021-11-02 (Actual)

PRIMARY OUTCOMES:
ASAS 20 responder | Week 16
  clinical response to treatment was assessed according to ASAS20 criteria. ASAS20 responder had improvement of 20% or more and absolute improvement of at least 1 units (on a scale of 0 [least] to 10 [worst]) from Baseline in at least 3 of the following 4 domains, with absence of deterioration (worsening of at least 20% an absolute Worsening of at least 1 unit) in the potential remaining domain: Patient's Global Assessment of Disease Activity; Total Back Pain visual analog scale (VAS); Function (Bath Ankylosing Spondylitis Functional Index (BASFI)); and Inflammation (mean of 2 morning stiffness-related Bath Ankylosing Spondylitis Disease Activity Index [BASDAI] scores

SECONDARY OUTCOMES:
ASAS 40 responder | Week 2, 4, 8, 12, 16, 20, 24
  Number of Participants Who Achieved ASAS40，ASAS40 responder had improvement of 40% or more and absolute improvement of at least 2 units (scale of 0 [least] to 10 [worst]) from Baseline in at least 3 of the following 4 domains, with no deterioration in the potential remaining domain: Patient's Global Assessment of Disease Activity; Total Back Pain visual analog scale (VAS); Function (Bath Ankylosing Spondylitis Functional Index (BASFI)); and Inflammation (mean of 2 morning stiffness-related Bath Ankylosing Spondylitis Disease Activity Index [BASDAI] scores)
ASAS 5/6 responder | Week 12, 16, 24
  Number of Participants Who Achieved ASAS5/6，ASAS 5/6 responder had improvement of 20% or more) from Baseline in at least 5 of the following 6 domains: Patient's Global Assessment of Disease Activity; Total Back Pain visual analog scale (VAS); Function (Bath Ankylosing Spondylitis Functional Index (BASFI)); and Inflammation (mean of 2 morning stiffness-related Bath Ankylosing Spondylitis Disease Activity Index [BASDAI] scores); Spinal Mobility (BASFI); Acute phase reactant (CRP)
Mean Change Bath Ankylosing Spondylitis Metrology Index (BASMI) Score | Week 2, 4, 8, 12, 16, 20, 24
  BASMI measures the range of motion based on five clinical measurements: 1) cervical rotation, 2) tragus to wall distance, 3) lumbar side flexion, 4) lumbar flexion (modified Schober's) and 5) intermalleolar distance. BASMI 0 = indicates mild disease involvement, 1 = moderate disease, and 2 = severe disease involvement. The results for cervical rotation and lumbar side flexion are the means of the left and right measurements. Scoring range 0-10. The higher the BASMI score, the more severe was the subject's limitation of movement
17. Change From Baseline in Bath Ankylosing Spondylitis Disease Activity Index (BASDAI) | Week 2, 4, 8, 12, 16, 20, 24
  The BASDAI consists of a 1 through 10 scale (1 being no problem and 10 being the worst problem), which was used to answer 6 questions pertaining to the 5 major symptoms of AS: Fatigue, Spinal pain, Joint pain / swelling, areas of localized tenderness (called enthesitis, or inflammation of insertion sites of tendons and ligaments), morning stiffness duration, and morning stiffness severity. The physician will globally assess the subject's current disease state
Magnetic Resonance Imaging (MRI) Inflammatory Scores | Week 16, 24
  The study used MRI with fat-saturating techniques such as short tau inversion recovery (STIR) to look for the presence of bone marrow edema. The Berlin modification of ASspiMRI-a (ASspiMRI-a) scoring technique assesses inflammation in each of the 23 disc vertebral units (DVU), capturing edema and erosion. Scores for each DVU range from 0-3 (0=normal; 1=minor bone marrow edema (less than25% of DVU; 3=severe bone marrow edema (more that 50% of DVU). The composite score ranges from 0 to 69, with higher scores indicating more severe inflammation
Number of adverse events to measure Safety of subcutaneously administered GR1501 | to Week 24
  Safety of GR1501 s.c. injection will be documented as numbers of adverse event

OTHER OUTCOMES:
ADA | Week 0, 2, 4, 16, 24
  Immunogenicity index (GR1501 antibody)
IL-17A | Week 0, 4, 16
  Peripheral blood IL-17A level

CONTACTS AND LOCATIONS:
Overall Officials: Xiaofeng Zeng, PHD, Principal Investigator — chairman
Locations (1):
- Peking Union Medical College Hospital, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No
within six months after the trail complete